CLINICAL TRIAL: NCT02383693
Title: Maintenance rTMS for Treatment-resistant Depression (TRD): a One-year Double Blind Controlled Study
Acronym: TMS/DEP
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre hospitalier de Ville-Evrard, France (Other)
Responsible Party: Principal Investigator, René BENADHIRA, MD, Centre hospitalier de Ville-Evrard, France
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007-A00244-49
Record Dates: First submitted 2015-02-24; First posted 2015-03-09 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Major Depressive Disorder
Keywords: depression; Repetitive Transcranial Magnetic Stimulation; tolerability; efficiency; TMS; refractory
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- repetitive transcranial magnetic stimulation (Active Comparator): Repetitive Transcranial Magnetic Stimulation (rTMS) Treatment 5 days/week for up to 4 weeks
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Sham comparator (Sham Comparator): Placebo Comparator: Placebo Treatment 5 days/week for up to 4 weeks
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Repetitive Transcranial Magnetic Stimulation
  Other Names: TMS

SUMMARY:
number of center : 1

* duration of study : 24 months
* recruitement time : 23 months
* Aim :Principal

Evaluate the interest of maintenance rTMS in a one-year double blind randomized controlled study for TRD patients.

Secondary

Evaluate the impact of rTMS on cognitive functions.

DETAILED DESCRIPTION:
The study involves 40 TRD patients in a single site trial which consisted of two phases: an acute phase (phase I) in which all the participants receive active high-frequency stimulation during 4 blocks of five consecutive working days (Monday to Friday) in an open-label design and a maintenance phase (phase II) in which responders (> 49% HDRS-17 reduction from baseline) at the end of the phase I are randomized in two arms with sham or active high-frequency rTMS maintenance treatment for the eleven following months. The rhythm of rTMS sessions in this maintenance phase is gradually reduced as follows: 3 sessions per week for 2 weeks, 2 session per week for the 2 following weeks, 1 session per week the third (M3) and fourth month (M4) and then 1 session every fortnight the last eight months (M5 to M12).

ELIGIBILITY:
Inclusion Criteria:

* TRD stage I Thase-Rush
* HDRS + or = 18
* Patients age 18 to 70 years.
* Negative pregnancy test and contraception for women.
* Informed Consent

Exclusion Criteria:

* Patient was treated with mood stabilizer in the previous week
* Other disorder on axis I of the DSM IV than depressive disorder.
* Patient with an addiction problem other than tobacco and caféine
* antécedent of Epilepsy ,other neurological pathology and intra cranial metal diapositive or pacemaker
* Previous history of head trauma the previous two years.
* intracranial hypertension.
* not affiliated to the social security Patient
* patient under constraint hospitalisation
* Under legal protection measure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
'Hamilton depression rating scale (HDRS) | one years
  The efficacy variables included the HDRS-17 item scores, the CGI changes, the Visual Analog Scale (VAS), the Beck Depression Inventory (BDI) and the Hospital Anxiety Depression (HAD).
  The subjective assessment performed with the VAS consisted of a 100-mm horizontal line oriented with anchors placed at both poles for reassured, sadness, anxiety, and relief. The patients are asked to mark a spot along this line that best indicated the magnitude of their state for each item.

CONTACTS AND LOCATIONS:
Overall Officials: Rene BENADHIRA, MD, Principal Investigator — E.P.S ville Evrard
Locations (1):
- Unité de Recherche Clinique, Neuilly-sur-Marne, Île-de-France Region, France